CLINICAL TRIAL: NCT05101044
Title: Improving Retention in Care for Persons With HIV Who Use Substances by Increasing Acceptance and Reducing Stigma (Open Trial)
Brief Title: Open Trial to Improve Retention in Care for Persons With HIV Who Use Substances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: The Miriam Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2104002974; R34DA053738 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Substance Use Disorders; Hiv
Keywords: Acceptance and commitment therapy; Acceptance-based behavioral therapy; Behavioral intervention; Acceptability and feasibility; Stigma
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Social Stigma | interventions — Methods

STUDY DESIGN:
Intervention Model Description: An uncontrolled open trial approach will be used in which all participants receive the ABBT intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance-based Behavioral Therapy (ABBT) Intervention (Experimental): All recruited individuals will receive ABBT intervention. ABBT involves 2 sessions delivered within about a week of each other, consisting of a 20-25 minute session 1, and a 10 minute session 2.
  Interventions: Behavioral: Acceptance-based Behavioral Therapy (ABBT) Intervention

INTERVENTIONS:
Behavioral: Acceptance-based Behavioral Therapy (ABBT) Intervention — This acceptance-based behavioral therapy (ABBT) intervention intends to enhance retention in HIV care for people who use substances by targeting stigma. ABBT promotes an accepting stance towards life's challenges and encourages participants to thoughtfully disclose the serostatus and/or substance abuse problems as a behavioral step towards challenging stigmatization fears. The central hypothesis is that increased tolerance of stigmatization, facilitated through increased acceptance of HIV status and substance use behaviors, will increase PWH's longitudinal commitment to care.

SUMMARY:
The open trial will examine the feasibility and acceptability of a brief, empirically-supported acceptance-based behavioral therapy intervention to promote retention in care for out-of-care people with HIV who use substances.

DETAILED DESCRIPTION:
The proposed study will adapt a brief, 2-session acceptance-based behavioral therapy (ABBT) intervention to help people with HIV (PWH) who use substances tolerate fears of stigmatization, increase acceptance of HIV status and substance use problems, and increase engagement in care. By conducting an open trial with 15 adults recruited from an HIV primary medical care clinic, the study will focus on the feasibility of recruiting out-of-care PWH and determine the acceptability of the refined ABBT protocol.

ELIGIBILITY:
Inclusion Criteria:

1. HIV+
2. Meet DSM-5 criteria for one or more of the following substance use disorders, at any severity level: cocaine, methamphetamine, and/or opioid
3. ≥18 years old
4. Poorly retained in care, defined as no attended medical appointment in the past 9 months
5. Able to speak and read English at a level sufficient to complete the study procedures
6. Have telephone access

Exclusion Criteria:

(a) Patients who are cognitively impaired, which will be determined by chart review during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ) | 1 month
  The Client Satisfaction Questionnaire is a self-report measure of patient satisfaction with treatment. The total score will be used and ranges from 8 to 32 with increased scores indicating greater satisfaction with treatment.

SECONDARY OUTCOMES:
Participant Retention Rate Across Intervention Sessions | Baseline and 1 month
  The investigators will examine the percent of participants that complete all intervention sessions.
Participant Retention Rate for Follow Up Assessments | Baseline and 1 month
  The investigators will examine the percent of participants that complete the 1-month follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Moitra, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - The Miriam Hospital, Providence, Rhode Island
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No